CLINICAL TRIAL: NCT01866618
Title: Natural Cycle In Vitro Fertilization
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-2013-01
Record Dates: First submitted 2013-05-20; First posted 2013-05-31 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Natural Cycle in Vitro Fertilization (IVF)
Keywords: Natural; IVF Cycle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Natural IVF Cycle: All patients will undergo a natural IVF cycle using trigger shots of Leuprolide Acetate(Lupron) and human chorionic gonadotropin (hCG) to ensure the patient surges.

SUMMARY:
Natural IVF study patients will undergo an IVF cycle with trigger shots of Lupron & hCG. Patients will not be given any other stimulating medications during the cycle. They will have 2 uterine aspirations and an endometrial biopsy at designated times. The first uterine aspiration will be randomized to one of four days (day before retrieval, day of retrieval, day after retrieval or 2 days after retrieval). The second uterine aspiration and endometrial biopsy will be performed 6 days after retrieval. Any embryo(s) obtained will be biopsied for Comprehensive Chromosome Screening (CCS) and frozen for use in a subsequent thaw cycle.

ELIGIBILITY:
Inclusion Criteria:

* Ovulatory cycles every 39 days or less (natural cycle IVF cannot be performed in someone who does not have cycles)
* Must be RMANJ patient and have completed all diagnostic screening at one of our RMANJ locations. All diagnostic screening is NOT covered under the study and must be completed prior to being allowed to start the study cycle.

Exclusion Criteria:

* Prior enrollment/attempt in this study
* Requirement for surgical sperm extraction
* Inability to assess ovaries via transvaginal ultrasound
* Inability to tolerate vaginal examination

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile patients
Sampling Method: Non-Probability Sample
Enrollment: 524 (Actual)
Dates: Start 2013-04; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Endometrial Changes | 1 Year
  To examine the endometrium within the natural cycle in order to accurately characterize the differences in multiple aspects of endocrine and paracrine hormonal activity, the transcriptome of cells influencing oocyte maturation and changes in the endometrium.

SECONDARY OUTCOMES:
Aneuploidy Rates | 1 Year
  To examine aneuploidy rates in embryos from natural IVF cycles.

OTHER OUTCOMES:
Temporal Embryonic Development | 1 Year
  To examine the parameters of temporal embryonic development and the transcriptome of granulosa cells and follicular fluid. The embryos will be graded at standard time points to determine whether there are differences in in vitro development. Granulosa cells and follicular fluid will undergo gene expression analysis and compared to the gene expression profiles found in those specimens in stimulated cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, M.D., HCLD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

REFERENCES:
- [Derived] Hong KH, Franasiak JM, Werner MM, Patounakis G, Juneau CR, Forman EJ, Scott RT Jr. Embryonic aneuploidy rates are equivalent in natural cycles and gonadotropin-stimulated cycles. Fertil Steril. 2019 Oct;112(4):670-676. doi: 10.1016/j.fertnstert.2019.05.039. PMID 31561871